CLINICAL TRIAL: NCT06941753
Title: Effectiveness of Off-script Diagnosis & Differential Diagnosis (D&D) Training in Improving Residents' Competence in Acute Ischemic Stroke Diagnosis and Treatment
Brief Title: Off-script Diagnosis & Differential Diagnosis (D&D) Training and Residents' Stroke Knowledge
Acronym: CAST-AIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CAST-AIS2025
Record Dates: First submitted 2025-04-15; First posted 2025-04-24 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-04

CONDITIONS: Stroke, Acute; Educational Problems; Clinical Course
Keywords: resident; stroke education
MeSH Terms: conditions — Stroke; Disease Progression | interventions — Fumigant 93

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Off-script D&D training group (Experimental): Off-script D&D training is required within 72 hours after randomization.
  Interventions: Other: Off-script diagnosis & differential diagnosis (D&D) training
- No-Intervention Control Group (No Intervention): Off-script D&D training is not required within 72 hours after randomization.

INTERVENTIONS:
Other: Off-script diagnosis & differential diagnosis (D&D) training — 1. Training Timeline: Must be completed within 72 hours post-randomization; Requires standardized structured off-script D&D analysis.
  2. Structured Analysis Framework: 1)Epidemiology: Incidence, mortality, and disability rates; 2) Etiologic Classification: TOAST classification system; 3) Vascular Mechanisms: Culprit vessel, vascular territory, pathophysiology; 4) Differential Diagnosis: Stroke mimics and stroke subtype differentiation; 5) Acute Management: Hyperacute interventions (thrombolysis/EVT), secondary prevention strategies, and evidence-based case analysis; 6) Patient Education: Stroke prevention education for patients/public; 7) Research Gaps: Current limitations and future directions.
  3. Presentation Requirements: 1)Mandatory off-script delivery (no prepared text); 2) Time limit: 15+3 minutes for complete analysis.
  Arms: Off-script D&D training group

SUMMARY:
This study is a single-center, randomized, open-label, controlled, endpoint-blinded study to assess the effect of off-script diagnosis & differential diagnosis (D&D) training in improving the residents' knowledge of acute ischemic stroke in China. The investigators will enroll 22 residents and assess the score of mASMaQ 30 days after randomization.

DETAILED DESCRIPTION:
Ischemic stroke is characterized by high incidence and disability rates, with a critical time window for reperfusion therapy, necessitating prompt recognition, diagnosis, and treatment by frontline physicians. In clinical practice, residents across all specialties may encounter acute ischemic stroke (AIS) patients in emergency departments, outpatient clinics, or inpatient wards. However, many residents face challenges in managing AIS cases, often leading to missed diagnoses, treatment delays, and non-adherence to clinical guidelines. A primary contributing factor is their insufficient mastery of key AIS management principles and inability to effectively apply stroke knowledge in clinical contexts.

Enhancing residents' AIS management competence represents a significant challenge in stroke education. Traditional "Initial Progress Note" training overemphasizes comprehensive differential diagnoses, with most residents relying on scripted presentations. The actual clinical application of stroke knowledge remains uncertain. This study aims to evaluate whether off-script diagnosis & differential diagnosis (D&D) training (i.e., "Structured off-script D&D") can significantly improve residents' AIS management knowledge.

The investigators will enroll 22 neurology residents and randomly assign them to two groups: the off-script diagnosis & differential diagnosis (D&D) training group (n=11) and a blank control group (n=11). The modified Acute Stroke Management Questionnaire (mASMaQ) will be used to assess residents' AIS knowledge 30 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Residents (physicians in postgraduate training).
2. Currently in neurology wards
3. Managing acute ischemic stroke (AIS) patients, defined as: 1)Time from onset to randomization ≤ 2 weeks; 2) If onset time is unknown, the last known well time is considered the onset time.
4. Signed informed consent

Exclusion Criteria:

1. Managing asymptomatic ischemic stroke patients.
2. Residents who are currently participating or have participated in another interventional ischemic stroke training program within the past 3 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
mASMaQ | 30 days
  Modified Acute Stroke Management Questionnaire (mASMaQ), with a range of 33-165 scores. Higher scores indicate superior acute ischemic stroke management knowledge.
  Blinded Assessment Protocol:1) Participant Requirements: Strict 10-minute time limit for independent completion; External references are prohibited; 2) Assessment Supervision: certified neurologists as proctors, who are blinded to group assignment throughout the trial. 3) Centralized Adjudication: based on participants' questionnaire responses.
  Note: Details of the modified ASMaQ has been on file with the ethics committee and cannot be changed. To prevent disclosure of the measures and bias in resident measurement, we do not disclose the scales until the trial is completed. Details of mASMaQ will be made public with the publication of the article.

SECONDARY OUTCOMES:
General stroke knowledge | 30 days
  Part of mASMaQ, with a range of 10-50. Higher scores indicate superior general stroke knowledge.
Hyperacute stroke management | 30 days
  Part of mASMaQ, with a range of 9-45. Higher scores indicate superior hyperacute stroke management knowledge.
Advanced stroke management | 30 days
  Part of mASMaQ, with a range of 14-70. Higher scores indicate superior advanced stroke management knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ni, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No